CLINICAL TRIAL: NCT07294703
Title: Genomic and Non-Genomic Factors Associated With Breast Cancer Risk Factors and Outcomes
Brief Title: Factors Associated With Breast Cancer Risks and Outcomes
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 25-335
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Memorial Sloan Kettering Cancer Center; 25-335
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with a suspicious breast finding or new breast cancer diagnosis: Participants with a suspicious breast finding who present to breast radiology at MSK for biopsy or a participants with a new breast cancer diagnosis who is a surgical candidate seen at MSK.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Complete surveys:
  * Baseline (within 6 months of enrollment)
  * 1st follow-up survey (approx. 6 months to 12 months)
  * 2nd follow-up survey and/or blood collection (approx. 3 years +/- 6 months)
  * 3rd follow-up survey and/or blood collection (approx. 5 years +/- 6 months)

SUMMARY:
The purpose of this study is to learn more about risks and outcomes of breast cancer in people with different backgrounds. Tissue and blood will be collected from participants for research purposes. Participants will complete questionnaires during their standard medical care. The study will not provide treatment for cancer or any other condition.

ELIGIBILITY:
Women 18 years and older who are patients with a suspicious breast finding who present to breast radiology at MSK for biopsy or any new breast cancer patient seen at MSK undergoing surgery.

Inclusion Criteria:

A patient cannot be considered eligible for this study unless the following conditions are met.

* Patients with a suspicious breast finding who present to breast radiology at MSK for biopsy or any new breast cancer patient who is a surgical candidate seen at MSK.
* Women 18 years of age and older are eligible to participate in the study.

Exclusion Criteria:

* Patients presenting to radiology for biopsy with a suspicious breast mass less than 1 cm will be considered ineligible.
* Patients presenting to clinic with microinvasion will be considered ineligible.
* Patients who are less than 18 years of age will be considered ineligible.
* Patients unable to complete the survey, including IDMC patients.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MSK research staff and/or treating clinicians will identify participants (anyone meeting inclusion criteria listed above) prior to or during their regularly scheduled visits (Breast radiology at time of initial biopsy, Surgery clinic visit, Medical Oncology clinic visit). A member of the MSK study team will approach the participants either in person or remotely to explain details of the study and answer any questions.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2031-12-08 (Estimated); Study Completion 2031-12-08 (Estimated)

PRIMARY OUTCOMES:
Recurrence Free Survival/RFS | 5 years
  RFS as defined by the STEEP 2.0 guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Neha Goel, MD, MPH, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Cancer Center Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activites), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activites), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made following one year after publication and for up to 36 months later. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org